CLINICAL TRIAL: NCT07201441
Title: The Impact of Intelligent Nursing Based on Health Cloud Platform on Active Health Management of Urostomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023KY816
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): On the basis of routine nursing, the intelligent cloud platform management mode is added.
  Interventions: Behavioral: Smart Nursing Based on the Health Cloud Platform
- Control Group (Active Comparator): Implement routine nursing.
  Interventions: Behavioral: Smart Nursing Based on the Health Cloud Platform

INTERVENTIONS:
Behavioral: Smart Nursing Based on the Health Cloud Platform — On the day of surgery, ensure that the patient or their family members have followed the hospital's official account and bound the patient's information. Through the intelligent cloud platform on the mobile device, they can query the patient's inpatient information, such as examination reports and details of inpatient expenses, and also consult and communicate about the patient's condition.

SUMMARY:
Research data show that the incidence of bladder tumors in China ranks first among malignant tumors of the urinary system and is on the rise . Muscle - invasive bladder tumor is a fatal malignant tumor, and radical cystectomy with urinary diversion is the main treatment method . After urinary diversion, patients rely on urostomy for urination for life, unable to control urine at will, and need to wear ostomy bags for life, resulting in self - image disorder. Urostomy brings a lot of troubles to patients and their families, increases the economic burden, especially makes young patients feel anxious about life, lose confidence in the future, and causes great psychological pressure . Due to the strong professionalism of stoma care, with the improvement of medical technology, the average hospital stay of patients after surgery is shortened, resulting in patients not fully mastering the knowledge and skills of urostomy care at the time of discharge, and their self - care ability is at a low level. They are prone to various health problems, which directly affects the quality of life of patients and their families .

Health is an inevitable requirement for the all - around development of people. The "Healthy China 2030" Plan Outline emphasizes the concept of proactive health. Proactive health refers to long - term, continuous and dynamic tracking of an individual's behavior system, identification and assessment of one's own state, evolution direction and degree, selection of various elements of lifestyle as the main means, giving full play to one's subjective initiative, and conducting controllable interventions on human behavior to improve health behaviors. In 2017, the Ministry of Science and Technology issued a notice officially including proactive health in the special plan. The concept of proactive health management has become an important part of realizing the Healthy China strategy.

DETAILED DESCRIPTION:
Proactive health management mainly promotes health through five dimensions: Dimension 1: Improve "proactive health management literacy", Dimension 2: Accurately predict "health risks", Dimension 3: Intelligently warn of "health events", Dimension 4: Effectively intervene in "health outcomes", Dimension 5: Comprehensively improve "health level". Proactive health is needed for healthy people, and proactive health management is even more important for patients. As a special group in society, urostomy patients who face many health problems after discharge need proactive health management even more, as well as the care of their families and society and postoperative rehabilitation guidance .

Traditional post - discharge follow - up methods are time - consuming and energy - consuming, difficult to carry out fully, with a high rate of lost to follow - up and a high incidence of complications . Patients urgently need to solve new problems that occur after discharge. Guo Cheng et al. expounded on relevant suggestions for public hospitals to carry out medical science popularization work in the era of proactive health. As one of the first pilot provinces for "Internet + Nursing" in the country, our hospital responded to the national call and actively launched online nursing information services. The information platform providing online information services is a network virtual platform based on Internet technology with functions of information storage, management, sharing and processing. Our department, based on the hospital's health cloud platform for smart nursing services, shares the patient medical records in the hospital information system, records the information of urostomy patients, regularly pushes personalized health education to patients, regularly assesses patients' stoma care ability, and provides timely evaluation and feedback. At the same time, patients can solve problems through the graphic transmission or telephone consultation on the platform, promoting patients' participation in proactive health management.

At present, the research and practice of continuous nursing abroad have reached a mature stage, mainly including pre - discharge and post - discharge. Before discharge, senior clinical nurses ensure that patients receive appropriate continuous nursing through formulating comprehensive discharge plans. After discharge, community medical staff provide high - quality continuous services to patients . Sun V et al. created a stoma patient self - management program based on telehealth. This program carried out continuous nursing for enterostomy patients by establishing electronic health records, holding video conferences and transmitting graphics and texts.

In China, continuous nursing methods mostly rely on QQ（ Quick Query）, WeChat（ We Chat ） and video, pictures and text to promote postoperative rehabilitation. Mobile phone applications (APPs) based on the Internet, with the characteristics of high informatization, low cost, high speed and meeting individual needs, have become the main form of mobile medicine at present. Ji ping Zhu et al. carried out narrative follow - up nursing services for urostomy patients after discharge using the "Cloud Clinic" APP, reducing patients' postoperative anxiety, improving patients' ability to care for stomas and patient satisfaction. Actively responding to the call of the National Health Commission to carry out "Internet + Nursing Services", Wen et al. constructed an informatized management system for enterostomy patients' nursing based on the hospital information system, achieving the dynamics and comprehensiveness of medical and nursing information records. At the same time, it also provided patients with continuous nursing services such as online consultation and follow - up, but it still cannot achieve data communication between the internal and external networks.

The future development trend is to realize data sharing on the patient informatization management platform, which is convenient for medical staff to query and manage patient information, provides convenience for health consultation of stoma patients, ensures that patients receive timely attention and rehabilitation guidance after discharge, improves patients' self - care ability, reduces the incidence of complications, and improves patients' quality of life.

This study has been supported by the Medical and Health Research Project of Zhejiang Province (No. 2023KY816).

ELIGIBILITY:
Inclusion Criteria:

* Those with clear consciousness, distinct self - expression and without mental abnormalities.

Individuals whose age is between 18 and 80 years old (inclusive), and whose self - care ability (Barthel Index) score is greater than 90 points.

Those who are clearly aware of the diagnosis and have undergone total cystectomy with urostomy.

Patients without depression. Patients or their family members are able to use WeChat. Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients with tumor metastasis or combined with other tumors. Those with visual impairment. Vulnerable groups, including patients with mental illnesses, those with cognitive impairment, critically ill patients, minors, pregnant women, illiterate people, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Urostomy Self - care Score Urostomy Self - care Score Urostomy Self - care Score | The 1st, 3rd, and 6th months after surgery
  Developed by Kristensen , it includes 2 dimensions and 7 items. Each item is divided into 4 levels, scored from 0 to 3 points, with a total score ranging from 0 to 21 points. The higher the score, the higher the patient's self - care level. In 2014, Fu Suliang translated this scale into Chinese and tested its reliability and validity. The content validity index of the Chinese version of the Urostomy Self - care Scale is 0.952, and the Cronbach α coefficient is 0.88. It is suitable for measuring the self - care ability of patients with urostomy.

SECONDARY OUTCOMES:
Anxiety State Score | The 1st, 3rd, and 6th months after surgery
  The Self - Rating Anxiety Scale (SAS) is adopted: Developed by Zung in 1971, it is a self - rating scale containing 20 items with 4 - level scoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang, China